CLINICAL TRIAL: NCT07198113
Title: Clinical Outcomes of Medications Post Anti-TNF: Researching Effectiveness in Pediatric IBD
Brief Title: COMPARE - Pediatric Inflammatory Bowel Disease (PIBD)
Acronym: COMPARE
Status: Not yet recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 25-2019; Pro00118431 (Other: Duke University Health System IRB)
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis, Pediatric; Inflammatory Bowel Diseases; Crohn Disease
Keywords: Ulcerative colitis, pediatric; Inflammatory bowel disease, pediatric; IBD; CD; UC; PIBD; Pediatrics; Children; Anti-TNF; Vedolizumab; Ustekinumab; Risankizumab; Guselkumab; Mirikizumab; Tofacitinib; Upadacitinib; Patient-reported outcomes (PROs); Tumor necrosis factor antagonists; IL-23 agent; PCORI; PCORnet; DCRI; Duke; UNC; University of North Carolina; Observational cohort; Anti-tumor necrosis factor (TNF) refractory; Comparative Effectiveness Research (CER); COMPARE
MeSH Terms: conditions — Pediatric ulcerative colitis; Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Optional biospecimens will be collected throughout this study for future, unspecified research and may include blood, saliva, stool, and tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Children with Crohn's disease (CD): Pediatric CD patients initiating non-anti-TNF biologics and small molecules that are FDA-approved for adult populations
- Children with Ulcerative Colitis (UC): Pediatric UC patients initiating non-anti-TNF biologics and small molecules that are FDA-approved for adult populations
- Retrospective Safety Analysis: Retrospective cohort focused on the long-term safety of non-anti-TNF biologics and small molecules that are FDA-approved for adult populations in for CD and or UC. Electronic health record (EHR) data (retrospective cohort) will be collected from medical charts and EHRs at participating institutions.

SUMMARY:
The purpose of the study is to compare the clinical effectiveness and safety of newer inflammatory bowel disease (IBD) medications in anti-tumor necrosis factor (TNF) refractory patients with pediatric IBD (PIBD). Refractory means that there was no clinical response to anti-tumor necrosis factor (TNF) drugs or that the if there was a response, it is no longer present. The main question this study aims to answer is:

Are the newer medications used to treat IBD just as safe and effective for treating IBD in children.

Participants will already be taking these newer medications as assigned by their regular health care provider.Participants' care will be managed by their regular healthcare provider as part of usual (standard) care for those with PIBD. While taking these medications, participants will be asked to answer questions about their symptoms and health periodically over the course of the study.

DETAILED DESCRIPTION:
COMPARE is a multi-center, observational cohort study that includes both prospective and retrospective components and two patient population cohorts-Crohn's disease (CD) and ulcerative colitis (UC). The study will recruit pediatric IBD patients initiating non-anti-TNF biologics and small molecules that are FDA-approved for adult populations. The primary analyses in each cohort will compare the two most frequently used classes, with all IL-23 agents analyzed as a single class. Secondary comparisons will be conducted for any classes initiated by at least 50 participants. The investigators will also perform a retrospective cohort study using EHR data extracted from participating sites.

IL-23 agents could be any of the following medications:

* Vedolizumab (trade name Entyvio™)
* Ustekinumab (trade name Stelara™)
* Risankizumab (trade name Skyrizi™)
* Guselkumab (trade name Tremfya™)
* Mirikizumab (trade name Omvoh™)
* Tofacitinib (trade name Xeljanz™)
* Upadacitinib (trade name Rinvoq™)

While taking these medications, participants (or parent/caregiver proxies) will complete patient-reported outcome surveys (PROS) at baseline, every 2 months for the first 12 months, and every 6 months during the 2nd and 3rd years of follow-up. The surveys will collect information about the participants' general health and well-being while taking these medications.

Clinical follow-up will occur in the context of routine care (e.g., clinic visits, telehealth encounters) for a minimum of 1-year and up to 3 years after the index date, regardless of whether the participant remains on the index treatment. The study anticipates relatively standard follow-up for each participant, based on best clinical practice, while allowing for natural variation.

The study will collect data abstracted from the medical charts of enrolled participants. Baseline data, including potential confounders described in the statistical analysis plan, will be collected by sites upon participant enrollment or shortly thereafter. Follow-up data will be collected with each outpatient gastrointestinal (GI) visit, hospitalization, surgery, colonoscopy, imaging test (MRI, CT, intestinal ultrasound), laboratory test (unless electronically captured), IBD medication change, and adverse events.

In addition, structured electronic health record (EHR) data on enrolled participants will be extracted using automated queries utilizing the PCORnet® PCORnet Common Data Model (CDM) to supplement case report forms. EHR data extraction will include laboratory values, anthropometrics, emergency department (ED) visits (and diagnosis codes), hospitalizations (and diagnosis codes), antibiotic/antiviral prescriptions, encounter dates, and diagnosis codes for events of special interest (e.g., infections, malignancy, blood clots).

The study will collect and record adverse events from participants and their caregivers, as well as via regular EHR queries using the PCORnet® CDM.

Prospective enrollment is expected to take approximately 36 months with a minimum follow-up of 12 months for each participant (maximum of 36 months).

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years at study enrollment
* Diagnosis of CD, UC, or IBD-U by standard diagnostic criteria
* Prior non-response or loss of response to one or more anti-TNF agents
* Planning to initiate treatment with any of the following comparator agents: vedolizumab (α4β7 integrin antibody), ustekinumab (anti-IL-12/23 antibody), risankizumab, guselkumab, or mirikizumab, (IL-23 inhibitors), tofacitinib (JAK inhibitor), and upadacitinib (JAK inhibitor). Biosimilars or generic medications for any of the above will also be allowed and handled/analyzed in an identical manner to originators.
* Ability to provide child assent, if required per regulatory or local institutional guidelines, and parental informed consent in English or Spanish

Exclusion Criteria:

* Plans to change care to a different center within 1 year
* Prior use of a comparator agent (i.e., only patients starting their first comparator medication as monotherapy following anti-TNF will be eligible)
* Contraindication to any of the treatments under investigation
* Patients with UC or IBD-U who have undergone colectomy
* Patients with current ostomy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Crohn's disease (CD) or ulcerative colitis (UC) whose disease is refractory to anti-TNF therapy
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Measure of Crohn's disease (CD) impact on patients' daily lives (TUMMY CD) | Baseline, months 2, 4, 6, 8, 10, 12, 18, 24, 30, 36
  The TUMMY CD patient reported outcome (PRO) has been developed and is undergoing validation. For our CD cohort, we will collect data on both the TUMMY-CD and the PROMIS IBD PROs. If TUMMY-CD is proven to be a reliable and valid PRO by the time of our data analysis, we will utilize this as our primary PRO. Otherwise, we will rely on PROMIS IBD PROs. Change will be calculated as the difference between baseline and post-baseline scores, with higher scores reflecting greater symptom severity.
Measures of ulcerative colitis (UC) impact on patients' daily lives (TUMMY UC) | Baseline, months 2, 4, 6, 8, 10, 12, 18, 24, 30, 36
  Description: The TUMMY UC patient reported outcome (PRO) is a validated patient-reported outcome tool designed to assess gastrointestinal symptom burden in children and adolescents with ulcerative colitis (UC). Change will be calculated as the difference between baseline and post-baseline scores, with higher scores reflecting greater symptom severity. Scores range from 0 to 114 with higher values indicating greater symptom burden.
PROMIS Symptom Measure of Irritable Bowel Disease (IBD) | Baseline, months 2, 4, 6, 8, 10, 12, 18, 24, 30, 36
  NIH Patient Reported Outcome Measurement Information System (PROMIS) symptoms scale is a disease-specific PRO. Prior validation of the PROMIS IBD measure has demonstrated acceptable internal consistency (Cronbach's alpha of 0.74), as well as discriminative and known groups validity. The PROMIS IBD symptom score has been standardized such that a T score of 50 represents the median score in the reference pediatric IBD population. T scores range from 40 to 80 with higher scores indicating higher symptom burden and a minimal clinically important difference (MCID) of 5. We will not use the PROMIS IBD for measure of UC
Change in Pediatric PROMIS® Patient-Reported Outcome (PRO) Pain Interference Score for Crohn's Disease and Ulcerative Colitis (CD and UC) | Baseline, months 6, 12, 18, 24, 30, 36
  Pediatric Patient Reported Outcome Measurement Information System (PROMIS) assesses domains relevant to children and adolescents with CD and UC and their reported pain score. PROMIS Pediatric PROs domains have been standardized such that a T score of 50 represents the median score in the reference pediatric IBD population with higher scores indicating higher symptom burden and minimal clinically important difference (MCID) of 5.
Change in Pediatric PROMIS® Fatigue Score for Crohn's Disease and Ulcerative Colitis (CD and UC) | Baseline, months 6, 12, 18, 24, 30, 36
  Pediatric Patient Reported Outcome Measurement Information System (PROMIS) assesses domains relevant to children and adolescents with CD and UC and their reported fatigue score. PROMIS Pediatric PROs domains have been standardized such that a T score of 50 represents the median score in the reference pediatric IBD population with higher scores indicating higher symptom burden and minimal clinically important difference (MCID) of 5.
Change in Pediatric PROMIS® Anxiety Score for Crohn's Disease and Ulcerative Colitis (CD and UC) | Baseline, months 6, 12, 18, 24, 30, 36
  Pediatric Patient Reported Outcome Measurement Information System (PROMIS) assesses domains relevant to children and adolescents with CD and UC and their reported anxiety score. PROMIS Pediatric PROs domains have been standardized such that a T score of 50 represents the median score in the reference pediatric IBD population with higher scores indicating higher symptom burden and minimal clinically important difference (MCID) of 5.
Change in Pediatric PROMIS® Depression Score for Crohn's Disease and Ulcerative Colitis (CD and UC) | Baseline, months 6, 12, 18, 24, 30, 36
  Pediatric Patient Reported Outcome Measurement Information System (PROMIS) assesses domains relevant to children and adolescents with CD and UC and their reported depression score. PROMIS Pediatric PROs domains have been standardized such that a T score of 50 represents the median score in the reference pediatric IBD population with higher scores indicating higher symptom burden and minimal clinically important difference (MCID) of 5.
Change in sPCDAI Score for Crohn's Disease | Each clinic visit (baseline through follow-up, up to 3 years)
  The short Pediatric Crohn's Disease Activity Index (sPCDAI) is a validated tool to assess disease activity in children with Crohn's disease. It is based on clinical symptoms, physical examination findings, and laboratory values. Scores range from 0 to 90, with higher scores indicating greater disease activity. The outcome will be measured as the mean change in sPCDAI score from baseline to follow-up. T Scores ≤15 indicate remission, > 15-29 mild disease and ≥30 indicate moderate to severe disease
Change in Pediatric Ulcerative Colitis Activity Index (PUCAI) Score | Each clinic visit (baseline through follow-up, up to 3 years)
  The Pediatric Ulcerative Colitis Index (PUCAI) is a patient-centered, 6-item measure assessing abdominal pain, stool characteristics, and patient functioning. Scores ranging from 0 - 85 with higher scores indicate more disease activity. A cut-point of <10 indicates remission, ≥10 to 34 mild disease, ≥35-65 moderate disease, and ≥65 severe disease. Response is defined as a reduction of ≥ 20 points.

SECONDARY OUTCOMES:
Change in Fecal Calprotectin Concentration (CD and UC) | 12 months after after taking prescribed medication for CD or UC
  Fecal calprotectin is a noninvasive biomarker of intestinal inflammation. Stool samples will be collected at baseline and follow-up visits. Calprotectin concentration will be measured in micrograms per gram (µg/g) of stool. The outcome will be measured as the mean change in fecal calprotectin from baseline to follow-up. Higher values indicate greater intestinal inflammation. A threshold of < 150 μg/g will be used to define remission.
Number of Participants Experiencing Adverse Events (CD and UC) | After medication administration and every 3 months, up to 3 years
  Safety will be assessed by collecting and monitoring all adverse events (AEs) and serious adverse events (SAEs). Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), where applicable. The outcome will be summarized as the number of participants experiencing AE/SAE of grade 2 or higher.
Proportion of Participants Experiencing Adverse Events (CD and UC) | After medication administration and every 3 months, up to 3 years
  Safety will be assessed by collecting and monitoring all adverse events (AEs) and serious adverse events (SAEs). Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), where applicable. The outcome will be summarized as the proportion of participants experiencing AE/SAE of grade 2 or higher.
Exploration of Heterogeneity of Treatment Effects (HTE) Across Clinical Subgroups (CD and UC) | Baseline through follow -up for up to 3 years
  Heterogeneity of treatment effects (HTE) will be evaluated per baseline phenotype query that will run against the electronic health record (EHR) at sites. Treatment effects will be estimated within each subgroup (CD and UC) and compared to assess differential response patterns. This analysis is intended to identify variability in treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Kappelman, MD, Principal Investigator — Universty of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Health System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.